CLINICAL TRIAL: NCT07200401
Title: A Feasibility Study to Explore the Safety, Acceptability and Potential Cost Effectiveness of Self-swabbing at Home to Obtain Usable Surgical Wound Culture Swabs
Brief Title: Exploring if Patients Can Safely and Easily Swab Their Own Surgical Wounds at Home
Acronym: TREASURE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Collaborators: University of Nottingham (Other); Liverpool Heart and Chest Hospital NHS Foundation Trust (Other); Health Innovation East Midlands (Unknown); Birmingham Community Healthcare NHS (Other Government); University Hospitals Sussex NHS Foundation (Unknown); Centre for Healthcare Equipment and Technology Adoption (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IRAS 356847
Record Dates: First submitted 2025-08-12; First posted 2025-10-01 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-09

CONDITIONS: Cardiac Surgery; Infection, Soft Tissue; Wound Healing; Swabs; Self Management
Keywords: swab; wound; self-swab; home swabbing; surgical; surgery; infection
MeSH Terms: conditions — Soft Tissue Infections; Wounds and Injuries; Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Self-Swabbing Group (Experimental): ≥18 years old with median sternotomies (central wounds) after cardiac surgery will be drawn from two hospital sites
  Interventions: Procedure: Self-swabbing of surgical wound

INTERVENTIONS:
Procedure: Self-swabbing of surgical wound — Participants will perform self-swabbing of their surgical wound under observation by a research practitioner via secure video call.

SUMMARY:
The goal of this observational feasibility study is to learn if patients can safely, acceptably, and effectively collect their own wound swabs at home to detect clinically significant organisms in adults aged 18 and over who have had cardiac surgery via median sternotomy (central chest wound). Participants will be recruited from two sites: Harefield Hospital (Guy's and St Thomas' NHS Foundation Trust, London) and the Royal Sussex County Hospital (University Hospitals Sussex, Brighton).

The main questions it aims to answer are:

* Can home-based patient self-swabbing of surgical wounds provide swabs of sufficient quality for microbiological testing?
* Is self-swabbing at home safe and acceptable to patients following cardiac surgery?
* Could this approach be a cost-effective way to monitor for surgical wound infections?

Participants will:

* Receive a co-designed self-swabbing instruction pack, created in collaboration with a patient and public working group and clinical experts.
* Be observed via Microsoft Teams by a research practitioner while self-swabbing (or having their carer do so) to assess usability and adherence to instructions.
* Participate in a brief interview to share their experiences and feedback on the instructions and swabbing process.
* Send completed swabs to the hospital laboratory for analysis to determine the usability and timeliness of the samples.

ELIGIBILITY:
Inclusion Criteria:

* Feasibility Study

  * Cardiac surgery ≥18 years old patients with a central chest wound, where the wound is a closed wound - assessed by the research nurse
  * Patients having elective or urgent surgery
  * Patients who have been discharged home or to a care home
  * Willing and able to provide written informed consent prior to participation in the clinical investigation.
  * Willing and able to comply with all study related procedures, with or without digital resource/internet access.

Exclusion Criteria:

* Feasibility Study

  * Cardiac surgery patients with open wounds extending beyond skin level, or where deep tissue, organs or implants are visible, wounds with constant or heavy discharge of fluid, wounds leaking pus at the time of the video consultation.
  * Patients having emergency or salvage surgery
  * Patients still in hospital
  * Patients with a dressing covering their wound at the time of the video consultation.
  * Congenital or acquired immunodeficiency, bone marrow disease, diabetes, autoimmune conditions requiring immunosuppressive treatment, any immunosuppressive medication at the time of consent or within the last 4 weeks before consent.
  * Undergoing active cancer treatment at time of consent/ or planning to start cancer treatment within the study period or completed cancer treatment within the last 4 weeks of the study commencing.
  * Patients who lack capacity to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-01-06 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants who successfully perform self-swabbing at home | months 7-11
  The proportion of participants who successfully perform self-swabbing at home approximately two weeks post-discharge, with the swab sample delivered to the laboratory within 24 hours and deemed viable for laboratory analysis.
Participant ratings on the acceptability of the swabbing process | months 7-11
  assessed through participant interviews
Adherence to the swabbing protocol | months 7-11
  Number of participants who adhere to the swabbing protocol. Evaluated during observations conducted at the time of swabbing and during follow-up interview
Adverse events during the swabbing process | months 7-11
  Adverse events during the swabbing process evaluated during observations conducted at the time of swabbing and during follow-up interviews

SECONDARY OUTCOMES:
Participant ratings on the acceptability of the swabbing instructions | Immediately after the self-swabbing process during participant interviews (months 7-11)
  Acceptability of the swabbing instructions will be measured through participant interviews.
Participant ratings on the acceptability of the swabbing kit | Immediately after the self-swabbing process during participant interviews (months 7-11)
  Acceptability of the swabbing kit will be measured through participant interviews
Transport Time taken for swabs to reach the laboratory | months 7-11
  Measured in hours, collected during laboratory processing
Number of usable swabs (viable for analysis) | months 7-11
  Measured during laboratory processing
Recruitment and retention rates | months 7-11
  To be measured continuously during the trial to inform the design of a larger trial
Patient demographics distribution | months 7-11
  To be measured continuously during the trial to inform the design of a larger trial
New swabbing at home pathway | months 7-11

CONTACTS AND LOCATIONS:
Overall Officials: Sunil Bhudia, Principal Investigator — Royal Brompton and Harefield Hospitals, part of Guy's and St Thomas' NHS Foundation Trust (GSTFT); Ishtiaq Ahmed, Principal Investigator — University Hospitals Sussex NHS Foundation Trust
Locations (2):
- United Kingdom (2):
  - Royal Sussex County Hospital, Brighton
  - Harefield Hospital, Harefield

IPD SHARING:
Plan to Share IPD: Yes
On completion of the study, anonymised quantitative data from the interviews and anonymised themed analysis of qualitative data from the interviews will be stored in and made publicly available through the University of Nottingham data repository (https://rdmc.nottingham.ac.uk/)
URL: https://rdmc.nottingham.ac.uk/

REFERENCES:
- [Background] Census - Office for National Statistics (ons.gov.uk) Accessed 07/07/2024
- [Background] Tanner J, Brierley Jones L, Westwood N, Rochon M, Wloch C, Rogers LJ, Vaja R, Dearling J, Wilson K, Harrington P, Brown CS, Murphy G. Exploratory study of patients' and carers' preferences for postdischarge surgical wound monitoring using survey and interviews. BMJ Open. 2025 Jan 25;15(1):e087320. doi: 10.1136/bmjopen-2024-087320. PMID 39863412
- [Background] M. Rochon (2023) Surgical Site Infection surveillance: Time for a new agenda? Society of Tissue Viability: Advances in surgical wound management and reducing surgical site infection.(SSI) https://societyoftissueviability.org/whats-on/advances-in-surgical-wound-management-and-reducingsurgical-site-infection-ssi/
- [Background] Atchison C, Pristera P, Cooper E, Papageorgiou V, Redd R, Piggin M, Flower B, Fontana G, Satkunarajah S, Ashrafian H, Lawrence-Jones A, Naar L, Chigwende J, Gibbard S, Riley S, Darzi A, Elliott P, Ashby D, Barclay W, Cooke GS, Ward H. Usability and Acceptability of Home-based Self-testing for Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) Antibodies for Population Surveillance. Clin Infect Dis. 2021 May 4;72(9):e384-e393. doi: 10.1093/cid/ciaa1178. PMID 32785665
- [Background] Rochon M, Jawarchan A, Ingusan S, Cariaga K and Morais C. 'Project ID007672: Clinical audit of patient-reported antibiotics for wound problems following surgery and review of alternative strategies'. 25/02/2023. Unpublished.
- [Background] NHS England. Delivering a net zero National Health Service. Greener NHS " Delivering a 'Net Zero' National Health Service (england.nhs.uk) Accessed 27/02/2024
- [Background] NHS England. The NHS Long Term Plan. NHS England " The NHS Long Term Plan. Accessed 27/02/2024
- [Background] Royal College of General Practitioners. RCGP response to the Antimicrobial resistance national action plan: Call for evidence. Accessed 29/02/2024
- [Background] Antimicrobial Resistance Collaborators. Global burden of bacterial antimicrobial resistance in 2019: a systematic analysis. Lancet. 2022 Feb 12;399(10325):629-655. doi: 10.1016/S0140-6736(21)02724-0. Epub 2022 Jan 19. PMID 35065702
- [Background] GIRFT 2019 GIRFT National Survey April 2019 Layout 1 (gettingitrightfirsttime.co.uk)
- [Background] Tanner J, Padley W, Davey S, Murphy K, Brown B. Patient narratives of surgical site infection: implications for practice. J Hosp Infect. 2013 Jan;83(1):41-5. doi: 10.1016/j.jhin.2012.07.025. Epub 2012 Oct 22. PMID 23088921
- [Background] Cardiothoracic Interdisciplinary Research Network. Electronic address: CIRNetwork@outlook.com; National Cardiac Benchmarking Collaborative; Public Health England; Cardiothoracic Interdisciplinary Research Network. National survey of variations in practice in the prevention of surgical site infections in adult cardiac surgery, United Kingdom and Republic of Ireland. J Hosp Infect. 2020 Dec;106(4):812-819. doi: 10.1016/j.jhin.2020.09.016. Epub 2020 Sep 19. PMID 32956785
- [Background] UKHSA Surveillance of surgical site infections in NHS hospitals in England: April 2022 to March 2023. London UKHSA 2023
- [Background] Rochon M, Cariaga K, Sa F, et al. 2023 The unrecognised burden of post-discharge antibiotic consumption for surgical wounds. Abstract. The 37TH EACTS Annual Meeting 4- 7 October 2023, Vienna, Austria. Programme (y-congress.com)
- [Background] Research reveals levels of inappropriate prescriptions in England - GOV.UK (www.gov.uk)
- [Background] Woelber E, Schrick EJ, Gessner BD, Evans HL. Proportion of Surgical Site Infections Occurring after Hospital Discharge: A Systematic Review. Surg Infect (Larchmt). 2016 Oct;17(5):510-9. doi: 10.1089/sur.2015.241. Epub 2016 Jul 27. PMID 27463235
- [Background] Wounds UK Prevention 2023 Identification and Management of Surgical Wound Dehiscence (SWD) SN23_CD_SWD_WUK-web.pdf (wounds-uk.com) Accessed 08/07/2024
- [Background] Han SM, Greenfield G, Majeed A, Hayhoe B. Impact of Remote Consultations on Antibiotic Prescribing in Primary Health Care: Systematic Review. J Med Internet Res. 2020 Nov 9;22(11):e23482. doi: 10.2196/23482. PMID 33031045
- [Derived] Rochon M, Tanner J, Cariaga K, Harris R, Wilson K, Newby C, Kariwo K, Sowole L, Bolton SJ, Bouttell J, Ahmed I. Is home-based self-swabbing feasible for postoperative wound culture after cardiac surgery? A multicentre mixed-methods feasibility study in the UK. BMJ Open. 2026 Feb 10;16(2):e112691. doi: 10.1136/bmjopen-2025-112691. PMID 41667168